CLINICAL TRIAL: NCT03387696
Title: Mucormycosis in ICU: A French Multicenter Cohort Study
Brief Title: Mucormycosis in ICU
Acronym: ZygoRéa
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: ZygoRea (38RC17.008)
Record Dates: First submitted 2017-12-01; First posted 2018-01-02 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Mucormycosis
Keywords: Mucormycosis; Intensive Care Medicine
MeSH Terms: conditions — Mucormycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mucormycosis is an invasive fungal infection affecting patients with various clinical conditions especially patients with heavy immunosuppression or patients with trauma or extensive burns.

ZygoRéa is a retrospective and multicentric French study aimed to evaluate survival of patients with mucormycosis admitted in ICU at day-28 after admission. This study will also try also to describe the epidemiology of patients admitted in ICU.

DETAILED DESCRIPTION:
Mucormycosis is an invasive fungal infection affecting patients with various clinical conditions especially patients with heavy immunosuppression or patients with trauma or extensive burns. The incidence of Mucormycosis is currently increasing reaching 7% of invasive fungal infections in some immunocompromised patients. Because of its aggressive nature, Mucormycosis is associated with poor survival and high morbidity ; mortality is estimated between 16% and 64% according to different retrospective studies. No study has ever evaluated prognosis of patients with mucormycosis admitted in intensive care units (ICU).

ZygoRéa is a retrospective and multicentric French study aimed to evaluate survival of patients with mucormycosis admitted in ICU at day-28 after admission. This study will also try also to describe the epidemiology of patients admitted in ICU and to evaluate the prognosis of different subgroups of patients according to :

* their clinical characteristics : demographic characteristics, clinical conditions and factors of immunosuppression
* the characteristics of the fungal infection
* the treatment strategy
* the severity of the initial illness, evaluated by severity scores

Twenty-one French ICU are currently including more than 45 patients.

ELIGIBILITY:
Inclusion Criteria:

* confirmed or suspected mucormycosis, based on international definition from EORTC/MSG
* patient hospitalized in intensive care unit during the 2008-2016 period
* Zygomycosis identification in at least 2 solids organs or identification in hemoculture

Exclusion Criteria:

* Age under 18 years old
* Patient under the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with mycormycosis hospitalized in intensive care unit during the 2008-2016 period
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Mortality at Day 28 | up to 28 days
  Mortality at Day 28 after ICU admission

SECONDARY OUTCOMES:
Mortality at Day 90 | up to 90 days
  Mortality at Day 90 after ICU admission
Mortality during the ICU stage | up to 28 days
  Mortality status (alive or dead) at the end of the ICU stage
Length stay in ICU | up to 28 days
  number of days in intensive care Unit
Length stay of hospitalization | up to 90 days
  number of days in hospital
Mortality during the hospitalization | up to 90 days
  Mortality status (alive or dead) at the end of the hospitalization
Prognostic criteria | up to 28 days
  Prognostic factors of mortality in intensive care units

CONTACTS AND LOCATIONS:
Locations (21):
- France (21):
  - Intensive Care Unit - Hospital Amiens, Amiens
  - Intensive Care Unit - Hospital Angers, Angers
  - Intensive Care Unit - Hospital Besançon, Besançon
  - Intensive Care Unit - Hospital Béthune, Béthune
  - Intensive Care Unit - Hospital Caen, Caen
  - Intensive Care Unit - Hospital Clermont-Ferrand, Clermont-Ferrand
  - Intensive Care Unit - Hospital Dijon, Dijon
  - Intensive Care Unit - Hospital Grenoble Alpes, Grenoble
  - Intensive Care Unit - Hospital Lille, Lille
  - Intensive Care Unit - Hospital Lyon, Lyon
  - Intensive Care Unit - Hospital Montpellier, Montpellier
  - Intensive Care Unit - Hospital Nantes, Nantes
  - Intensive Care Unit - Hospital l'Archet - Nice, Nice
  - Intensive Care Unit - Hospital Bichat, Paris
  - Intensive Care Unit - Hospital Saint Louis, Paris
  - Intensive Care Unit - Hospital Tenon, Paris
  - Intensive Care Unit - Hospital Poitiers, Poitiers
  - Intensive Care Unit - Hospital Rennes, Rennes
  - Intensive Care Unit - Hospital Rouen, Rouen
  - Intensive Care Unit - Hospital Saint Etienne, Saint-Etienne
  - Intensive Care Unit - Hospital Tours, Tours

IPD SHARING:
Plan to Share IPD: No